CLINICAL TRIAL: NCT06264154
Title: The Role of Flavor in the Substitutability of E-cigarettes for Combustible Cigarettes Among Persistent Smokers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Janet E. Audrain-McGovern, PhD, Professor, University of Pennsylvania
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UPCC 11023; R01CA287474-01 (NIH); 854051 (Other: University of Pennsylvania IRB Protocol Number)
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Smoking; Tobacco Use; Cigarette Smoking; E-Cig Use
MeSH Terms: conditions — Smoking; Tobacco Use; Cigarette Smoking; Vaping | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fruit-flavored E-cigarettes (Experimental): Participants randomized to fruit-flavored e-cigarettes will be provided with an e-cigarette device and be instructed to switch from smoking combustible cigarettes to using only the study provided e-cigarette device and fruit-flavored nicotine pods. Participants will be able to choose between blueberry or watermelon-flavored pods. They will receive their supply of nicotine pods in 7-day increments, based on baseline smoking behavior.
  Interventions: Other: E-cigarettes
- Tobacco-flavored E-cigarettes (Active Comparator): Participants randomized to tobacco-flavored e-cigarettes will be provided with an e-cigarette device and be instructed to switch from smoking combustible cigarettes to using only the study provided e-cigarette device and tobacco nicotine pods. Participants will receive their supply of nicotine pods in 7-day increments, based on baseline smoking behavior.
  Interventions: Other: E-cigarettes
- Menthol-flavored E-cigarettes (Active Comparator): Participants randomized to menthol-flavored e-cigarettes will be provided with an e-cigarette device and be instructed to switch from smoking combustible cigarettes to using only the study provided e-cigarette device and menthol nicotine pods. Participants will receive their supply of nicotine pods in 7-day increments, based on baseline smoking behavior.
  Interventions: Other: E-cigarettes

INTERVENTIONS:
Other: E-cigarettes — All participants are instructed to switch from smoking combustible cigarettes to using e-cigarettes for 6 weeks. Participants will receive an e-cigarette device and flavored nicotine pods according to their randomly assigned flavor.

SUMMARY:
This between-subjects study aims to evaluate the effect of flavor on initial and sustained switching from combustible cigarettes to e-cigarettes among 210 cigarette smokers. After measuring baseline cigarette smoking rate, participants will be randomized to a six-week regimen of fruit-flavored, tobacco-flavored, or menthol-flavored e-cigarettes and be instructed to switch (versus smoking cigarettes) over a 6-week period. Flavor-associated subjective reward and the reinforcing value of flavored e-cigarettes relative to combustible cigarettes will be assessed as mechanisms.

DETAILED DESCRIPTION:
The average smoker will attempt to quit smoking at least 30 times before abstaining for 12 months or longer. These attempts typically occur over decades of smoking, carcinogen and toxicant exposure, resulting in 480,000 deaths annually. As highlighted in the Surgeon General's Report, helping smokers who cannot quit smoking switch to less harmful non-combustible nicotine-containing products, such as e-cigarettes, has the potential to reduce this health burden dramatically. Substituting e-cigarettes for combustible cigarettes might only be possible for persistent smokers if e-cigarettes are accessible and appealing. Harm reduction proponents have advocated for the continued availability of e-cigarette flavors to appeal to and aid cigarette smokers unable to quit with traditional methods. Yet, there are no prospective studies of the effect of flavor on initial and sustained switching from combustible to electronic cigarettes. Converging laboratory, epidemiological, and clinical research suggests that fruit-flavored e-cigarettes with nicotine may be a viable substitute for combustible cigarettes among persistent smokers. The proposed study seeks to answer two novel questions relevant to public health and the regulation of e-cigarette flavoring. First, do persistent smokers substitute fruit-flavored e- cigarettes more readily than traditional-flavored e-cigarettes (tobacco or menthol) for combustible cigarettes? Second, are fruit-flavored e-cigarettes more rewarding and reinforcing than traditional-flavored e-cigarettes, and do these effects facilitate switching? The proposed research will fill these gaps in the evidence base by randomizing 210 persistent cigarette smokers to a six-week regimen of fruit-flavored (FF: watermelon and blueberry, n=70), tobacco-flavored (TF n=70) or menthol-flavored (MF n=70) e-cigarettes in a between-subjects design. Baseline smoking rate will be established during days 1-5. After biochemically verified overnight cigarette smoking abstinence, laboratory visits on days 6 and 7 will assess flavor-associated subjective reward and the reinforcing value of flavored e-cigarettes relative to combustible cigarettes. Participants will then switch from cigarette smoking to e-cigarette use for six weeks. Participants will collect spent cigarette filters daily to assess cigarettes smoked per day (cpd) if they smoke. The primary outcome measure is the longitudinal daily count of cigarettes from baseline to the end of the six-week switch period, with cigarettes per day at a 6-month follow-up as a secondary endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Able to communicate fluently in English (i.e. speaking, writing, and reading)
2. Male and female smokers who are > 21 years of age and self-report smoking at least 5 cigarettes (menthol and/or non-menthol) per day for at least the last 12 months
3. 5 or more failed quit attempts and the use of smoking cessation medication on at least one prior attempt.
4. Ever use of an e-cigarette
5. Have a carbon monoxide (CO) greater than 10 ppm
6. Not using any forms of nicotine regularly other than cigarettes
7. Be willing to switch to e-cigarettes for 6 weeks and use the assigned flavors
8. Plan to live in the area for the duration of the study
9. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the combined consent and HIPAA form.

Exclusion Criteria:

Smoking Behavior Regular use of nicotine-containing products other than cigarettes (e.g., chewing tobacco, snuff, snus, cigars, e-cigs, etc.). Regular e-cigarette use is defined as greater than 5 days/past 30 days

1. Participants agreeing to abstain from using nicotine-containing products other than cigarettes for the duration of the study will be considered eligible.
2. Current enrollment or plans to enroll in a smoking cessation program over the duration of the study.
3. Current use of smoking cessation medication
4. Provide a CO breath test reading less than 10 ppm at Intake.

Alcohol and Drug

1. History of substance abuse (other than nicotine dependence) in the past 12 months.
2. Current alcohol consumption that exceeds 20 standard drinks/week.
3. Current use of recreational drugs (other than nicotine and cannabis)
4. Breath alcohol reading (BrAC) greater than .000 at Intake.

Medical

1. Women, including all individuals assigned as "female" at birth, who are pregnant, breastfeeding, or planning a pregnancy over the duration of the study period.
2. Serious or unstable disease within the past year (e.g. cancer, heart disease). Applicable conditions will be evaluated on a case-by-case basis by the Principal Investigator.
3. Allergies to either propylene glycol or flavor additives

Psychiatric

1. Lifetime history of schizophrenia or psychosis.

General Exclusion

1. Past, current, anticipated, or pending enrollment in another research program over the study period that could potentially impact subject safety, study data, and/or the study design as determined by the Principal Investigator.
2. Any medical condition, illness, disorder, adverse event (AE), or concomitant medication that could compromise participant safety or significantly impact study performance as determined by the Principal Investigator. Subjects may be deemed ineligible for any of the aforementioned reasons at any point throughout the study, as well as during the initial telephone screen.
3. Significant non-compliance with protocol and/or study design as determined by the Principal Investigator and/o. Subjects may be deemed ineligible at any point throughout the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Cigarette Consumption | 42 days (days 8 - 49)
  The primary outcome is the longitudinal daily count of cigarettes from baseline to the end of the e-cigarette switch phase. Daily cigarette consumption will be determined by counting the daily spent cigarette filters returned for each of the 42 days (days 8 - 49).
Cigarette Smoking Behavior | 19 Weeks (Day 50-6-Month Follow-Up)
  Cigarette smoking behavior at the 6-month follow-up will serve as a secondary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Audrain-McGovern, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States